CLINICAL TRIAL: NCT06362473
Title: Lipid Transport Disorder Italian Genetic Record (LIPIGEN)
Acronym: LIPIGEN
Status: Recruiting | Type: Observational
Sponsor: Fondazione SISA (Societa Italiana per lo Studio della Arteriosclerosi) (Other)
Responsible Party: Sponsor
Other Study IDs: LIPIGEN-001
Record Dates: First submitted 2024-04-02; First posted 2024-04-12 (Actual); Last update posted 2024-04-12 (Actual); Status verified 2024-04

CONDITIONS: Familial Hypercholesterolemia; Genetic Disorder
Keywords: LIPIGEN; Familial Hypercholesterelomia; Genetic Dyslipidemia
MeSH Terms: conditions — Hyperlipoproteinemia Type II; Genetic Diseases, Inborn

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Lipid-lowering treatments

SUMMARY:
LIPIGEN is an observational study involving Italian physicians and researchers in the field of diseases related to blood lipid levels. This study aims to improve the diagnosis and treatment of people with familial dyslipidaemias, including very common conditions such as familial hypercholesterolaemia (FH) and less common ones such as familial chylomicronidaemic syndrome (FCS).

What does the study do?

It collects information on Italian patients with Familial Hypercholesterolaemia (FH), following them in their normal clinical examination without adding extra procedures.

It uses the data collected to further our understanding of diseases such as familial hypercholesterolaemia, examining how it is diagnosed clinically and by genetic testing, and evaluating the effectiveness of different treatments.

It seeks to identify the genetic mutations that cause familial hypercholesterolaemia and other dyslipidaemias, helping to choose the most effective treatments.

It evaluates the impact of long-term treatments and patient adherence to medication, as well as monitoring the incidence of cardiovascular events and other important outcomes.

Who can participate?

The study is aimed at people of all ages, from children to adults, with familial hypercholesterolaemia or other genetic dyslipidaemia.

More than 50 centres throughout Italy are involved, making the study accessible to many.

What does participation entail?

Participants will continue with their normal clinical practice.

Data such as family history, personal clinical findings and genetic information will be collected, without additional procedures.

For some, further evaluations, such as ultrasounds, may be required to better study their condition.

The LIPIGEN study not only helps to better understand diseases related to high cholesterol but also aims to improve patients' lives through more precise diagnosis and personalised treatments.

ELIGIBILITY:
Inclusion Criteria:

* Molecular or clinical diagnosis of genetic dyslipidemia
* Informed consent signed

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Subjects with molecular or clinical diagnosis of genetic dyslipidemia of any age or sex.
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2015-08-04 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Lipid profile of patients with genetic dyslipidemia | At baseline evaluation
  Lipid profile of patients with molecular or clinical diagnosis of genetic dyslipidemia:
  * LDL cholesterol (mg/dL)
  * Total cholesterol (mg/dL)
  * HDL cholesterol (mg/dL)
  * Triglycerides (mg/dL)
  * Lipoprotein (a) (mg/dL), if available
Genetic profile of patients with genetic dyslipidemia | At baseline evaluation
  Genetic profile of patients with molecular or clinical diagnosis of genetic dyslipidemia:
  * Prevalance (%) of patients with pathogenic/likely pathogenic variants on candidate genes
  * Prevalance (%) of patients with variants of uncertain significance (VUS) on candidate genes
  * Distribution (%) of more common variants

CONTACTS AND LOCATIONS:
Overall Officials: Alberico L Catapano, PhD, Study Chair — Fondazione S.I.S.A.
Locations (1):
- IRCCS Multimedica, Sesto San Giovanni, Milano, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Averna M, Cefalu AB, Casula M, Noto D, Arca M, Bertolini S, Calandra S, Catapano AL, Tarugi P; LIPIGEN Group. Familial hypercholesterolemia: The Italian Atherosclerosis Society Network (LIPIGEN). Atheroscler Suppl. 2017 Oct;29:11-16. doi: 10.1016/j.atherosclerosissup.2017.07.001. PMID 28965615